CLINICAL TRIAL: NCT04649853
Title: Wound Care and Pressure Injury Through the Continuum of Care
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Regional Medical Center of San Jose (Other)
Responsible Party: Principal Investigator, Charleen Singh, Director of Wound Care Services, Regional Medical Center of San Jose
Other Study IDs: 1267389
Record Dates: First submitted 2020-08-17; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Wound; Pressure Injury
MeSH Terms: conditions — Wounds and Injuries; Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acute Wounds: Patient with either traumatic or surgical wounds
- Chronic Wounds: Patient with chronic wounds either peripheral vascular disease related or surgical/traumatic wound
- Pressure Injuries Present on Admission: Patient admitted with one or more pressure injury of any stage on admission
  Interventions: Other: Standardized nursing care
- At Risk for Pressure Injury: Patient admitted with risk for pressure injury and has no pressure injuries at time of admission. Identified as at risk for based on mobility.
  Interventions: Other: Standardized nursing care

INTERVENTIONS:
Other: Standardized nursing care — All patients will receive standardized evidence based nursing care
  Groups: At Risk for Pressure Injury; Pressure Injuries Present on Admission

SUMMARY:
Our primary objective is to understand the impact of our quality improvement objectives on pressure injury and wound care outcomes. We will follow patients admitted to our facility who receive the standard of care for a up to a year. Patients to be followed will fall into one of four groups: acute wounds, chronic wounds, pressure injuries present at time of admission and at risk for pressure injuries.

DETAILED DESCRIPTION:
Overall Objective The main objective is to understand the impact of an evidence-based best practice model for wounds and pressure injuries that follows a patient through the continuum of care.

Specific Aims The specific aim is to measure the rates of healing using tissue analytics and the rates of pressure injuries.

The secondary aim measured is patients understanding of their health and the impact on their wound healing, prevention of wound re-opening and pressure injury.

Once we identify the rates we can translate the impact of rates into healthcare dollars and begin to understand the fiscal impact of evidence based practice.

BACKGROUND AND SIGNIFICANCE

Over the past decade researchers published the benefit of advanced wound care and the need to implement pressure injury prevention. To date there is very little literature connecting the acute care and post-acute care as a continuum by following a patient. Little is known about what the outcomes for wound care and pressure injury would be if a patient were followed through the trajectory of care. The medical home model suggests that placing the patient at the center of care is the best practice for best outcomes. However, at times in the hustle of the healthcare system the patient is lost. Implementing evidence-based best practice that follows the patient through the continuum of care is one approach to keeping the patient at the center of care. Currently wound care and pressure injury care or prevention is practiced in silos between acute-care and post-acute care. There is little literature that links the impact of continuing care throughout the continuum.

RESEARCH DESIGN AND METHODS Overview This quantitative study will utilize both primary and secondary data. The secondary data source will come from chart review and be the comparison group for outcomes. Patients will be enrolled upon admission as they are identified as meeting criteria, which includes either having a chronic wound that is not followed by a vascular team or an acute wound or a pressure injury. The fourth group of individuals to be enrolled into the study are those patients who are immobile and are expected to remain immobile at the time of discharge. Patients will be identified by admitting clinical staff and then enrolled and consented by the study coordinator or principal investigator. Once enrolled in the study, patients will have evidence based best practice interventions implemented based on their needs while in the acute care setting. For patients with wounds this will include that their cover dressing will be an antimicrobial foam bordered dressing that minimizes dressing changes. For immobile patients they will have the evidence based best practice pressure injury prevention bundle implemented. During the acute care admission, the patient will receive education regarding their wound care and or pressure injury prevention. Once the target post-admission site is identified, education for the caregiver at the receiving site will be provided. The patient will continue to be followed in the post-acute setting until the wound is healed or six months has passed on a weekly basis for a maximum of time frame of one year. The wounds will be measured weekly using tissue analytics. Re-education and coaching will be provided to the post-acute care facility. As patients are discharged from the study, they will be asked to complete an evaluation survey of their satisfaction with the care and the impact on their lives. The caregivers in the post-acute care will be asked to complete a survey to evaluate the education and support provided.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria includes:

* 18 years and older
* admitted into acute care with acute wound
* admitted with chronic wound
* admitted with pressure injury
* at risk for pressure injury

Exclusion Criteria:

* pregnant patients
* patients under 18
* known vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target study sample are adults who have either an acute wound, chronic wound, pressure injury or at risk for a pressure injury that are admitted to the acute care organization. The primary site is a community based acute-care organization. Patients will be identified upon admission.
Sampling Method: Probability Sample
Enrollment: 352 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The implementation of evidence-based best practice for wound care in the acute-care setting that is extended into post-acute care will improve outcomes. | 1 year
  Rate of wound healing
The implementation of an evidence based pressure injury prevention bundle in acute care that is extended into post-acute care will prevent pressure injuries in high-risk patients. | 1 year
  Number of individuals who are at risk to develop a pressure injury actually develop pressure injuries
The implementation of an evidence based pressure injury prevention bundle for patients with existing pressure injuries will prevent new pressure injuries from occurring | 1 year
  Measurement of occurrence of new pressure injuries for individuals with existing pressure injuries
The extension of a best practice prevention bundle implemented in acute-care and extending into post-acute care will reduce fiscal expenditure. | 1 year
  Comparison of number of individuals admitted from post acute with pressure injuries to acute acute after receiving education and the fiscal impact.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Thorpe, MSN, Study Chair — Regional Medical Center San Jose
Locations (1):
- Regional Medical Center San Jose, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data is coded and stored on the hospital password protected server. We don't plan to share the data at this time.

REFERENCES:
- [Result] Swietek KE, Domino ME, Beadles C, Ellis AR, Farley JF, Grove LR, Jackson C, DuBard CA. Do Medical Homes Improve Quality of Care for Persons with Multiple Chronic Conditions? Health Serv Res. 2018 Dec;53(6):4667-4681. doi: 10.1111/1475-6773.13024. Epub 2018 Aug 7. PMID 30088272
- [Result] Berkowitz SA, Terranova J, Hill C, Ajayi T, Linsky T, Tishler LW, DeWalt DA. Meal Delivery Programs Reduce The Use Of Costly Health Care In Dually Eligible Medicare And Medicaid Beneficiaries. Health Aff (Millwood). 2018 Apr;37(4):535-542. doi: 10.1377/hlthaff.2017.0999. PMID 29608345
- [Result] Van Eenoo L, van der Roest H, Onder G, Finne-Soveri H, Garms-Homolova V, Jonsson PV, Draisma S, van Hout H, Declercq A. Organizational home care models across Europe: A cross sectional study. Int J Nurs Stud. 2018 Jan;77:39-45. doi: 10.1016/j.ijnurstu.2017.09.013. Epub 2017 Sep 21. PMID 29032349
- [Result] Campbell Britton M, Petersen-Pickett J, Hodshon B, Chaudhry SI. Mapping the care transition from hospital to skilled nursing facility. J Eval Clin Pract. 2020 Jun;26(3):786-790. doi: 10.1111/jep.13238. Epub 2019 Jul 16. PMID 31309664
- [Result] Meehan R. Transitions From Acute Care to Long-Term Care: Evaluation of the Continued Access Model. J Appl Gerontol. 2019 Apr;38(4):510-529. doi: 10.1177/0733464817723565. Epub 2017 Aug 8. PMID 28786316
- [Result] Molloy MA, Cary MP Jr, Brennan-Cook J, Cantey DS, Tocchi C, Bailey DE Jr, Oermann MH. Preparing Clinicians for Transitioning Patients Across Care Settings and Into the Home Through Simulation. Home Healthc Now. 2018 Jul/Aug;36(4):225-231. doi: 10.1097/NHH.0000000000000667. PMID 29979303
- [Result] Nussbaum SR, Carter MJ, Fife CE, DaVanzo J, Haught R, Nusgart M, Cartwright D. An Economic Evaluation of the Impact, Cost, and Medicare Policy Implications of Chronic Nonhealing Wounds. Value Health. 2018 Jan;21(1):27-32. doi: 10.1016/j.jval.2017.07.007. Epub 2017 Sep 19. PMID 29304937
- [Result] Pal A, Goswami D, Cuellar HE, Castro B, Kuang S, Martinez RV. Early detection and monitoring of chronic wounds using low-cost, omniphobic paper-based smart bandages. Biosens Bioelectron. 2018 Oct 15;117:696-705. doi: 10.1016/j.bios.2018.06.060. Epub 2018 Jul 5. PMID 30014943
- [Result] Brain D, Tulleners R, Lee X, Cheng Q, Graves N, Pacella R. Cost-effectiveness analysis of an innovative model of care for chronic wounds patients. PLoS One. 2019 Mar 6;14(3):e0212366. doi: 10.1371/journal.pone.0212366. eCollection 2019. PMID 30840658
- [Result] Olsson M, Jarbrink K, Divakar U, Bajpai R, Upton Z, Schmidtchen A, Car J. The humanistic and economic burden of chronic wounds: A systematic review. Wound Repair Regen. 2019 Jan;27(1):114-125. doi: 10.1111/wrr.12683. Epub 2018 Dec 2. PMID 30362646
- [Result] Padula WV, Pronovost PJ, Makic MBF, Wald HL, Moran D, Mishra MK, Meltzer DO. Value of hospital resources for effective pressure injury prevention: a cost-effectiveness analysis. BMJ Qual Saf. 2019 Feb;28(2):132-141. doi: 10.1136/bmjqs-2017-007505. Epub 2018 Aug 10. PMID 30097490
- [Result] Cheng Q, Graves N, Pacella RE. Economic Evaluations of Guideline-Based Care for Chronic Wounds: a Systematic Review. Appl Health Econ Health Policy. 2018 Oct;16(5):633-651. doi: 10.1007/s40258-018-0403-9. PMID 29968020
- [Result] Kapp S, Miller C, Santamaria N. The quality of life of people who have chronic wounds and who self-treat. J Clin Nurs. 2018 Jan;27(1-2):182-192. doi: 10.1111/jocn.13870. Epub 2017 Aug 9. PMID 28493644
- [Result] Holscher CM, Hicks CW, Canner JK, Sherman RL, Malas MB, Black JH 3rd, Mathioudakis N, Abularrage CJ. Unplanned 30-day readmission in patients with diabetic foot wounds treated in a multidisciplinary setting. J Vasc Surg. 2018 Mar;67(3):876-886. doi: 10.1016/j.jvs.2017.07.131. Epub 2017 Oct 7. PMID 29017807
- [Result] Martinengo L, Olsson M, Bajpai R, Soljak M, Upton Z, Schmidtchen A, Car J, Jarbrink K. Prevalence of chronic wounds in the general population: systematic review and meta-analysis of observational studies. Ann Epidemiol. 2019 Jan;29:8-15. doi: 10.1016/j.annepidem.2018.10.005. Epub 2018 Nov 12. PMID 30497932
- [Result] Padula WV, Pronovost PJ. Addressing the multisectoral impact of pressure injuries in the USA, UK and abroad. BMJ Qual Saf. 2018 Mar;27(3):171-173. doi: 10.1136/bmjqs-2017-007021. Epub 2017 Sep 19. No abstract available. PMID 28928166
- [Result] Courvoisier DS, Righi L, Bene N, Rae AC, Chopard P. Variation in pressure ulcer prevalence and prevention in nursing homes: A multicenter study. Appl Nurs Res. 2018 Aug;42:45-50. doi: 10.1016/j.apnr.2018.06.001. Epub 2018 Jun 5. PMID 30029713
- [Result] Dreyfus J, Gayle J, Trueman P, Delhougne G, Siddiqui A. Assessment of Risk Factors Associated With Hospital-Acquired Pressure Injuries and Impact on Health Care Utilization and Cost Outcomes in US Hospitals. Am J Med Qual. 2018 Jul;33(4):348-358. doi: 10.1177/1062860617746741. Epub 2017 Dec 20. PMID 29262690